CLINICAL TRIAL: NCT04723069
Title: A Randomized, Double-blind, Positive-Controlled Study to Evaluate the Efficacy and Safety of Fuke Qianjin Capsule in Patients With Pelvic Inflammatory Diseases
Brief Title: Efficacy and Safety of Fuke Qianjin Capsule in Patients With Pelvic Inflammatory Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Zhuzhou Qianjin Pharmaceutical Co., Ltd., 801, Zhuzhou, China (Unknown); Center for bioequivalence studies and Clinical Research (CBSCR), ICCBS, University of Karachi (Unknown)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-007-TCM-FKQJ -2020
Record Dates: First submitted 2021-01-22; First posted 2021-01-25 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Pelvic Inflammatory Disease
Keywords: Triditional Chinese Medicine; Pelvic Inflammatory Disease (PID); Doxycycline Hyclate; Metronidazole
MeSH Terms: conditions — Pelvic Inflammatory Disease | interventions — Control Groups; Medicine, Chinese Traditional

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, positive control
Who Masked: Participant, Investigator
Masking Description: Participant and investigator both are blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fuke Qianjin capsule (Experimental): Metronidazole tablets + Doxycycline Hyclate tablets simulant are consecutively taken for 14 days, while the Fuke Qianjin capsule is consecutively taken for 28 days.
  Fuke Qianjin Capsules are taken as 2 capsules at a time, 3 times a day, orally after breakfast, lunch, and dinner, respectively; Metronidazole Tablets are taken as 2 tablets (0.2 g/tablet) at a time, twice a day, at the same time as breakfast and dinner, respectively; Doxycycline Hyclate Tablet simulants are taken as 1 tablet (0.1 g/tablet, Doxycycline Hyclate Tablet calculated as C22H24N2O8) at a time, twice a day, at the same time as breakfast and dinner, respectively.
  Interventions: Drug: Control Group
- Metronidazole tablets + Doxycycline hyclate tablets (Active Comparator): Metronidazole tablets + Doxycycline hyclate tablets are consecutively taken for 14 days, while Fuke Qianjin capsule simulation is consecutively taken for 28 days.
  Fuke Qianjin Capsules simulants are taken as 2 capsules at a time, 3 times a day, orally after breakfast, lunch and dinner, respectively; Metronidazole Tablets are taken as 2 tablets (0.2 g/tablet) at a time, twice a day, at the same time as breakfast and dinner, respectively; Doxycycline Hyclate Tablet simulants are taken as 1 tablet (0.1 g/tablet, Doxycycline Hyclate Tablet calculated as C22H24N2O8) at a time, twice a day, at the same time as breakfast and dinner, respectively.
  Interventions: Drug: Test Group

INTERVENTIONS:
Drug: Control Group — metronidazole tablets + doxycycline hyclate tablets, are consecutively taken for 14 days, while Fuke Qianjin capsule simulation is consecutively taken for 28 days.
  Other Names: Traditional Chinese Medicine (TCM)
  Arms: Fuke Qianjin capsule
Drug: Test Group — metronidazole tablets + doxycycline hyclate tablets simulant are consecutively taken for 14 days, while Fuke Qianjin capsule is consecutively taken for 28 days.
  Arms: Metronidazole tablets + Doxycycline hyclate tablets

SUMMARY:
Randomized, double blind and positive-controlled clinical trial to assess the efficacy and safety of Fuke Qianjin Capsule compared to Doxycycline Hyclate Tablet in patients with mild to medium PID and its sequalae.

DETAILED DESCRIPTION:
Study participants will be randomly assigned to Test or Control group and the following schedule will be followed

Test group: metronidazole tablets + doxycycline hyclate tablets simulant are consecutively taken for 14 days, while Fuke Qianjin capsule is consecutively taken for 28 days.

Control group: metronidazole tablets + doxycycline hyclate tablets, are consecutively taken for 14 days, while Fuke Qianjin capsule simulation is consecutively taken for 28 days.

Fuke Qianjin Capsules and their simulants are taken as 2 capsules at a time, 3 times a day, orally after breakfast, lunch and dinner, respectively; Metronidazole Tablets are taken as 2 tablets (0.2 g/tablet) at a time, twice a day, at the same time as breakfast and dinner, respectively; Doxycycline Hyclate Tablet and their simulants are taken as 1 tablet (0.1 g/tablet, Doxycycline Hyclate Tablet calculated as C22H24N2O8) at a time, twice a day, at the same time as breakfast and dinner, respectively.

Scoring pain, symptoms, local signs, routine leucorrhea, cervical secretions, gynaecological B-ultrasound will be examined before the enrollment and after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-55.
* History of sexual life.
* Consistent with the diagnosis of pelvic inflammatory disease.
* VAS score ≥4.
* Voluntarily participate in the clinical trial and signed the Informed Consent form obtained before any trial-related procedures are performed

Exclusion Criteria:

* Patients with severe pelvic inflammatory disease, or patients with dizziness, vomiting, high fever; pelvic abscess; fallopian tube ovarian abscess, etc.
* Absence of uterus.
* Patients with gynaecological tumors (uterine fibroids > 5 cm in diameter, submucosal fibroids), specific vaginitis, adenomyosis, endometriosis, pelvic venous stasis, tuberculous pelvic inflammatory disease, abnormal uterine bleeding, etc. confirmed by examination, and related symptoms caused by other diseases.
* Patients with serious primary diseases of the heart, liver, kidney, hematopoietic system and those who have an impact on clinical trial as judged by the investigator.
* Patients with neurological and psychiatric disorders and unable or unwilling to cooperate.
* Allergic (allergic to two or more substances) or allergic to the components of this medicine; Suspected or indeed history of allergy to tetracyclines.
* Pregnant and breastfeeding women.
* Treated with similar drugs in the past 2 weeks.
* Those who are participating in or have participated in other clinical trials in the past 3 months.
* Suspected or confirmed history of alcohol or drug abuse, or other lesions or conditions that may reduce the possibility or complicate enrolment according to the judgment of the investigator, such as frequent changes in work environment and unstable living environment, which may easily lead to loss of follow-up.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females with Pelvic inflammatory Disease are Eligible.
Enrollment: 198 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Improvement in Visual Analog Scale (VAS) for pain assessment | after 28 days of treatment
  Applying the Visual Analogue Scale (VAS) i.e. 0-10 Numeric Pain Intensity Scale on a 10 cm line segment the pain will be assessed as 0 is painless, 10 is extremely painful. Patients will mark in the corresponding position according to the degree of pain, and the researcher will give a specific score. The grading criteria of Pelvic pain with VAS score will be, normal: 0 cm; mild: 1-3 cm; moderate: 4-6 cm; severe: 7-10 cm.

SECONDARY OUTCOMES:
Assessment of changes in main clinical Symptom | after 28 days of treatment
  Main Clinical symptoms including Lower abdominal pain (Score 0 points: No Pain, 2 points: Mild, 4 points: Moderate and 6 points: Severe ), Lumbosacral pain (Score 0 points: No Pain, 2 points: Mild, 4 points: Moderate and 6 points: Severe ) and Yellow leucorrhea (Score 0 points: Normal, 2 points: light yellow, 4 points: yellow discharge and 6 points: Yellowish green as pus),
gynaecological B-ultrasound | after 28 days of treatment
  Change in the maximum area of pelvic effusion

OTHER OUTCOMES:
Labaratory Examination | at day 0, 14 and after 28 days of treatment
  Routine blood tests for liver function (alanine aminotransferase ALT, aspartate aminotransferase AST, γ-glutamyltransferase GGT, alkaline phosphatase ALP, total bilirubin T.BIL); Blood routine (WBC, RBC, HB, PLT, NEU%, LYM%, MONO%, EOS%); Urine routine (LEU, ERY, PRO, GLU, pH, KET); Liver function (AST, ALT, TBiL, ALP, GMT, LDH, AMS); Renal function (BUN, Cr, UA); Electrolytes(Na+, K+, Cl-, Ca+).
Vital signs examination | at day 0, 14 and after 28 days of treatment
  Blood Pressure Monitoring (Both systolic and diastolic), Body Temperature, Pulse rate, Respiratory Rate
Electrocardiogram | at day 0, 14 and after 28 days of treatment
  ECG evaluation for any abnormality

CONTACTS AND LOCATIONS:
Overall Officials: Professor Dr. Muhammad Raza Shah, Principal Investigator — Center for bioequivalence studies and Clinical Research (CBSCR), ICCBS, University of Karachi
Locations (1):
- Center for Bioequivalence Studies and Clinical Research (CBSCR), ICCBS, university of Karachi, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah MR, Khan SN, Fatima S, Yao L, Yuan H, Ullah S, Ainuddin J, Zeng C, Zheng Y, Sahar N, Anwar S, Zhu M, Ma C, Kumari K, Wang W, Liu R. A randomized, double-blind, positive-controlled, Phase-II clinical trial to evaluate efficacy and safety of Fuke Qianjin capsule in Pakistani patients with pelvic inflammatory disease. Front Pharmacol. 2024 Mar 22;15:1287321. doi: 10.3389/fphar.2024.1287321. eCollection 2024. PMID 38584600
- See also: The Clinical Effect of Fuke Qianjin Capsule on Chronic Pelvic Pain Caused by Pelvic Inflammation — https://clinicaltrials.gov/ct2/show/NCT03251560